CLINICAL TRIAL: NCT07033104
Title: Analgesic Effect of Adding Calcitonin to Bupivacaine in Transversalis Fascia Plane Block for Cesarean Section, A Prospective Randomized Study
Brief Title: Adding Calcitonin to Bupivacaine in Transversalis Fascia Plane Block for Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Abogabal, Marwa Abogabal, Tanta University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR1160
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Transversalis Fascia Plane Block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transversalis fascia plane block with bupivacaine (Active Comparator): us guided transversalis fascia plane block with bupivacaine
  Interventions: Other: us guided Transversalis fascia plane block
- Transversalis fascia plane block with calcitonin and bupivacaine (Active Comparator): us guided transvesalis fascia plane block with calcitonin and bupivacaine
  Interventions: Other: us guided Transversalis fascia plane block

INTERVENTIONS:
Other: us guided Transversalis fascia plane block — addition of calcitonin to pubivacaine

SUMMARY:
Evaluate calcitonin as an adjuvant to bupivacaine in ultrasound guided tansversalis fascia plane block

ELIGIBILITY:
Inclusion Criteria:

* female pt ASA2 scheduled for cs under spinal anesthesia

Exclusion Criteria:

* patient refusal ASAmore than 3 patients with pregnancy related disease emergency cs history of coagulopathy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
time to first rescue analgesia | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- tanta University hospital, Tanta, Gharbia Governorate, Egypt